CLINICAL TRIAL: NCT03224299
Title: Effectiveness of an Antimicrobial Agent for Preoperative Skin Preparation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MPS-16IPVFT05
Record Dates: First submitted 2017-07-10; First posted 2017-07-21 (Actual); Results first posted 2021-04-23 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-03

CONDITIONS: Preoperative Skin Preparation
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Investigational Product #1 (IP1) (Experimental): octenidine dihydrochloride in isopropyl alcohol in a single-use applicator - clear
  Interventions: Drug: OCT - clear
- Investigational Product #2 (IP2) (Experimental): octenidine dihydrochloride in isopropyl alcohol in a single-use applicator - tinted
  Interventions: Drug: OCT- tinted
- Active Control (Active Comparator): ChloraPrep® - Hi-Lite Orange® applicator
  Interventions: Other: ChloraPrep
- Negative Control (Placebo Comparator): sterile 0.9% saline applied with single use applicator
  Interventions: Other: Saline

INTERVENTIONS:
Drug: OCT - clear — Investigational Product #1: octenidine dihydrochloride in isopropyl alcohol in a single-use applicator - clear
  Arms: Investigational Product #1 (IP1)
Drug: OCT- tinted — Investigational product #2: octenidine dihydrochloride in isopropyl alcohol in a single-use applicator - tinted
  Arms: Investigational Product #2 (IP2)
Other: ChloraPrep — Active Control: ChloraPrep® - Hi-Lite Orange® applicator
  Arms: Active Control
Other: Saline — Negative Control: sterile 0.9% saline applied with single use applicator
  Arms: Negative Control

SUMMARY:
Objective of this study is to compare the antimicrobial properties of an investigational agent to an active control and a negative control when applied to specific body locations. Testing will be performed according to the procedures outlined in the Food and Drug Administration Tentative Final Monograph (TFM) for Effectiveness Testing of a Patient Preoperative Skin Preparation

ELIGIBILITY:
Inclusion Criteria:

* Subjects may be of either sex, at least 18 years of age and of any race.
* Subjects must be in good general health.
* Subjects must read and sign an Informed Consent Form, Authorization to Use and Disclose Protected Health Information Form, and the List of Restricted Products prior to participating in the study.
* Female subjects must complete a urine pregnancy test and have negative results documented before proceeding to treatment with test materials.
* All subjects must meet Screening Day microbial baseline requirements established by the sponsor.

Exclusion Criteria:

* Known allergies or sensitivities to sunscreens, deodorants, laundry detergents, fragrances, vinyl, latex (rubber), alcohols, soaps, metals, inks, dyes, tape adhesives, or to common antibacterial agents found in soaps, lotions, ointments, or particularly the active ingredients of the study product drug solutions.
* Exposure of test sites to strong detergents, solvents, or other irritants within the 14-day product-restriction period or during the test period.
* Exposure of test sites to antimicrobial agents, medicated soaps, medicated shampoos, or medicated lotions, use of biocide-treated pools or hot tubs, use of tanning beds, or sunbathing during the 14-day product-restriction period or during the test period.
* Wear fabric softener-, bug repellent-, or UV-treated clothing during the 14-day product-restriction period or during the test period.
* Use of systemic or topical antibiotic medications, steroid medications (other than for hormonal contraception or post-menopausal reasons), or any other product known to affect the normal microbial flora of the skin during the 14-day product-restriction period or during the test period.
* A medical diagnosis of a physical condition, such as a current or recent severe illness, mitral valve prolapse with a heart murmur, congenital heart disease, hepatitis B, hepatitis C, an organ transplant, ports, or an immunocompromised condition such as AIDS (or HIV positive), lupus, medicated diabetes (Type 1 or 2), ulcerative colitis, Crohn's disease, asthma requiring daily medication, fibromyalgia or multiple sclerosis (medicated).
* Any tattoos or scars within 2 inches of the test sites; skin blemishes or warts may be permissible with the specific approval of the Principal Investigator or consulting physician.
* Dermatoses, cuts, lesions, active skin rashes, scabs, breaks in the skin or other skin disorders within 6 inches, on, or around the test sites.
* A currently active skin disease or inflammatory skin condition (for example, contact dermatitis, psoriasis, eczema) anywhere on the body that, in the opinion of the Principal Investigator, would compromise subject safety or study integrity.
* Subjects who receive an irritation score of 1 (any redness, swelling, rash, or dryness present in any treatment area) for any individual skin condition prior to the Screening Day baseline or Treatment Day baseline sample collection.
* Participation in another clinical study in the past 30 days or current participation in another clinical study at time of signing informed consent.
* Showering, bathing, or swimming within the 72 hour period prior to sampling for baseline screening, the test day, or throughout the test period.
* Pregnancy, plans to become pregnant or impregnate a sexual partner within the pre-test and test periods of the study, or nursing a child. All female subjects will be required to complete a urine pregnancy test on the day of test material application, prior to treatment. Both gender of subjects must be willing to use an acceptable method of contraception to prevent pregnancy for at least 14 days immediately preceding Treatment Day and throughout the duration of the study.
* Any medical condition or use of any medications that, in the opinion of the Principal Investigator or Consulting Physician, would preclude participation.
* Unwillingness to fulfill the performance requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2017-06-21 (Actual); Primary Completion 2017-08-24 (Actual); Study Completion 2017-10-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - BioScience Laboratories, Bozeman, Montana
  - BioScience Laboratories, Butte, Montana

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Number of participants enrolled is 131. Each participant has up to 4 sites on their body treated with assigned products. Participants are treated bilaterally on the abdomen and/or groin based on passing screening criteria.
Groups:
- Number of Participants: Participants were treated with 2 of 4 study products (IP#1 [OCT/IPA-clear], IP#2 [OCT/IPA-tinted], AC [ChloraPrep Hi-Lite Orange], or NC [0.9% saline]), 1 on the left side of the body (abdomen and inguen received the same product) and 1 on the right (abdomen and inguen received the same product). Therefore, treatment groups are not discrete categories and cannot be described by treatment group.
- Number of Sites: Test sites on body
Period: Overall Study
Arm/Group | Number of Participants | Number of Sites
Started (Enrolled) | 131 | 424
Treated With IP#1 | 65 | 101
Treated With IP#2 | 66 | 107
Treated With AC | 66 | 110
Treated With NC | 65 | 106
Completed | 131 | 424
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants were treated with 2 of 4 study products (IP#1 [OCT/IPA-clear], IP#2 [OCT/IPA-tinted], AC [ChloraPrep Hi-Lite Orange], or NC [0.9% saline]), 1 on the left side of the body (abdomen and groin received the same product) and 1 on the right (abdomen and groin received the same product). Therefore, treatment groups are not discrete categories and cannot be displayed by treatment group.
Groups:
- Treated Subjects: All treated subjects
Arm/Group | Treated Subjects
Number analyzed (Participants) | 131
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 81
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 119
  Unknown or Not Reported | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 119
  More than one race | 0
  Unknown or Not Reported | 8
Region of Enrollment [Number; unit: participants]
  United States | 131

OUTCOME MEASURES:

1. Primary Outcome: Antimicrobial Activity of the Investigational Products Compared to Control.
Time Frame: 10 minutes
Population: Analysis only includes participants with required treatment day baseline bacterial counts at each anatomical site at baseline and non-missing data at 30 seconds and 10 minutes.
Measure: Mean (Standard Deviation); unit: log10 CFU/cm^2
Groups:
- Investigational Product #1: Octenidine dihydrochloride in isopropyl alcohol in a single-use applicator - clear
- Investigational Product #2: Octenidine dihydrochloride in isopropyl alcohol in a single-use applicator - tinted
Arm/Group | Investigational Product #1 | Investigational Product #2 | Active Control | Negative Control
Number analyzed (Participants) | 65 | 66 | 66 | 65
log10 CFU/cm^2
  Abdomen Baseline: number analyzed (Participants) | 38 | 44 | 47 | 47
  Abdomen Baseline | 3.85 (0.51) | 3.91 (0.52) | 3.87 (0.55) | 3.84 (0.55)
  Abdomen 30 seconds: number analyzed (Participants) | 38 | 44 | 46 | 47
  Abdomen 30 seconds | 0.98 (1.31) | 1.05 (1.23) | 1.34 (1.24) | 3.42 (0.72)
  Abdomen 10 minutes: number analyzed (Participants) | 38 | 44 | 47 | 47
  Abdomen 10 minutes | 1.20 (1.30) | 0.91 (1.15) | 1.08 (1.10) | 3.12 (0.87)
  Groin Baseline Groin Baseline: number analyzed (Participants) | 42 | 48 | 44 | 40
  Groin Baseline Groin Baseline | 6.03 (0.52) | 6.05 (0.59) | 6.03 (0.53) | 5.93 (0.50)
  Groin 30 seconds: number analyzed (Participants) | 42 | 47 | 43 | 40
  Groin 30 seconds | 2.91 (1.26) | 3.03 (1.16) | 3.05 (1.19) | 5.11 (0.41)
  Groin 10 minutes: number analyzed (Participants) | 42 | 48 | 44 | 40
  Groin 10 minutes | 2.37 (1.34) | 2.66 (1.37) | 2.66 (1.42) | 4.91 (0.43)
Statistical Analysis 1: Comparison: Investigational Product #1 vs Active Control; Abdomen 10 minutes Average treatment effect, calculated using a linear regression model for each body site, was used for primary analysis. In the model, the response was the post-treatment log10 bacterial counts and predictors were the treatment effect as a fixed effect and the pre-treatment log10 bacterial counts as a covariate; Test type: Non-Inferiority — Investigational product cannot be more than 0.05 log10 CFU/cm^2 less than the active control; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-0.44 to 0.69]
Statistical Analysis 2: Comparison: Investigational Product #1 vs Negative Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = 1.93, 95% CI 2-sided [1.36 to 2.49]
Statistical Analysis 3: Comparison: Investigational Product #2 vs Active Control; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — Investigational product cannot be more than 0.05 log10 CFU/cm^2 less than the active control; Mean Difference (Final Values) = -0.18, 95% CI 2-sided [-0.73 to 0.36]
Statistical Analysis 4: Comparison: Investigational Product #2 vs Negative Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = 2.23, 95% CI 2-sided [1.69 to 2.78]
Statistical Analysis 5: Comparison: Investigational Product #1 vs Active Control; Groin 10 minutes Average treatment effect, calculated using a linear regression model for each body site, was used for primary analysis. In the model, the response was the post-treatment log10 bacterial counts and predictors were the treatment effect as a fixed effect and the pre-treatment log10 bacterial counts as a covariate; Test type: Non-Inferiority — Investigational product cannot be more than 0.05 log10 CFU/cm^2 less than the active control; Mean Difference (Final Values) = -0.30, 95% CI 2-sided [-0.90 to 0.31]
Statistical Analysis 6: Comparison: Investigational Product #1 vs Negative Control; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; Mean Difference (Final Values) = 2.60, 95% CI 2-sided [1.98 to 3.22]
Statistical Analysis 7: Comparison: Investigational Product #2 vs Active Control; [analysis description as in outcome 1, analysis 5]; Test type: Non-Inferiority — Investigational product cannot be more than 0.05 log10 CFU/cm^2 less than the active control; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.61 to 0.57]
Statistical Analysis 8: Comparison: Investigational Product #2 vs Negative Control; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; Mean Difference (Final Values) = 2.33, 95% CI 2-sided [1.72 to 2.93]
Statistical Analysis 9: Comparison: Investigational Product #1 vs Active Control; Abdomen 30 seconds Average treatment effect, calculated using a linear regression model for each body site, was used for primary analysis. In the model, the response was the post-treatment log10 bacterial counts and predictors were the treatment effect as a fixed effect and the pre-treatment log10 bacterial counts as a covariate; Test type: Non-Inferiority — Investigational product cannot be more than 0.05 log10 CFU/cm^2 less than the active control; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-0.91 to 0.22]
Statistical Analysis 10: Comparison: Investigational Product #1 vs Negative Control; [analysis description as in outcome 1, analysis 9]; Test type: Superiority; Mean Difference (Final Values) = 2.45, 95% CI 2-sided [1.88 to 3.01]
Statistical Analysis 11: Comparison: Investigational Product #2 vs Active Control; [analysis description as in outcome 1, analysis 9]; Test type: Non-Inferiority — Investigational product cannot be more than 0.05 log10 CFU/cm^2 less than the active control; Mean Difference (Final Values) = -0.31, 95% CI 2-sided [-0.85 to 0.24]
Statistical Analysis 12: Comparison: Investigational Product #2 vs Negative Control; [analysis description as in outcome 1, analysis 9]; Test type: Superiority; Mean Difference (Final Values) = 2.41, 95% CI 2-sided [1.87 to 2.95]
Statistical Analysis 13: Comparison: Investigational Product #1 vs Active Control; Groin 30 seconds Average treatment effect, calculated using a linear regression model for each body site, was used for primary analysis. In the model, the response was the post-treatment log10 bacterial counts and predictors were the treatment effect as a fixed effect and the pre-treatment log10 bacterial counts as a covariate; Test type: Non-Inferiority — Investigational product cannot be more than 0.05 log10 CFU/cm^2 less than the active control; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.67 to 0.40]
Statistical Analysis 14: Comparison: Investigational Product #1 vs Negative Control; [analysis description as in outcome 1, analysis 13]; Test type: Superiority; Mean Difference (Final Values) = 2.25, 95% CI 2-sided [1.70 to 2.80]
Statistical Analysis 15: Comparison: Investigational Product #2 vs Active Control; [analysis description as in outcome 1, analysis 13]; Test type: Non-Inferiority — Investigational product cannot be more than 0.05 log10 CFU/cm^2 less than the active control; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.56 to 0.48]
Statistical Analysis 16: Comparison: Investigational Product #2 vs Negative Control; [analysis description as in outcome 1, analysis 13]; Test type: Superiority; Mean Difference (Final Values) = 2.15, 95% CI 2-sided [1.62 to 2.68]

2. Secondary Outcome: Responder Rate at 6 Hours Post-application
Description: Number of participants with bacterial reduction greater than or equal to baseline (0)
Time Frame: 6 hours
Population: Analysis only includes participants with required treatment day baseline bacterial counts at each anatomical site at baseline and non-missing data at 6 hours
Measure: Count of Participants; unit: Participants
Groups:
- IP#1: Investigational Product #1 (IP1) Octenidine dihydrochloride in isopropyl alcohol in a single-use applicator - clear
- IP#2: Investigational Product #2 (IP2) Octenidine dihydrochloride in isopropyl alcohol in a single-use applicator - tinted
- Active Control: Active Control (AC) - ChloraPrep® - Hi-Lite Orange® applicator
- Negative Control: Negative Control (NC) - Sterile 0.9% saline applied with single use applicator
Arm/Group | IP#1 | IP#2 | Active Control | Negative Control
Number analyzed (Participants) | 65 | 66 | 66 | 65
Participants
  Abdomen: number analyzed (Participants) | 38 | 44 | 47 | 47
  Abdomen | 37 | 43 | 47 | 42
  Inguen: number analyzed (Participants) | 42 | 48 | 44 | 40
  Inguen | 42 | 48 | 44 | 40

ADVERSE EVENTS:
Time Frame: 6 hours
Arm/Group | IP#1 | IP#2 | Active Control | Negative Control
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/66 | 0/66 | 0/65
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/66 | 0/66 | 0/65
Other Adverse Events (participants affected / at risk) | 0/65 | 0/66 | 0/66 | 0/65

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-04-19): https://cdn.clinicaltrials.gov/large-docs/99/NCT03224299/Prot_001.pdf
  • Statistical Analysis Plan (2017-08-02): https://cdn.clinicaltrials.gov/large-docs/99/NCT03224299/SAP_002.pdf